CLINICAL TRIAL: NCT00879333
Title: A Randomized, Double-blind, Multi-center Phase III Study Comparing Everolimus (RAD001) Plus Best Supportive Care Versus Placebo Plus Best Supportive Care in Patients With Advanced Gastric Cancer After Progression on 1 or 2 Prior Systemic Chemotherapy
Brief Title: Safety and Efficacy of RAD001 (Everolimus) Monotherapy Plus Best Supportive Care in Patients With Advanced Gastric Cancer (AGC)
Acronym: GRANITE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRAD001R2301; 2008-006544-20 (EudraCT Number)
Record Dates: First submitted 2009-04-08; First posted 2009-04-10 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Gastric Cancer
Keywords: Gastric cancer,; advanced gastric cancer,; stomach neoplasm,; stomach disease,; adenocarcinoma of stomach,; GI neoplasm
MeSH Terms: conditions — Stomach Neoplasms; Stomach Diseases; Digestive System Neoplasms | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus + BSC (Experimental): All patients were randomized to receive everolimus + BSC. All patients orally took two 5 mg tablets of everolimus once daily. Therefore, all patients in the everolimus arm took a total daily dose of 10 mg. Best supportive care was in accordance with the local practice of an individual institution or center, and specifically excluded anti-cancer treatments.
  Interventions: Drug: Everolimus; Drug: Best Supportive Care (BSC)
- Placebo + BSC (Placebo Comparator): All patients were randomized to receive placebo + BSC. All patients orally took two 5 mg tablets of matching placebo once daily. Therefore, all patients in the placebo receive matching tablets of total daily dose of 10 mg. Best supportive care was in accordance with the local practice of an individual institution or center, and specifically excluded anti-cancer treatments.
  Interventions: Drug: Everolimus placebo; Drug: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Everolimus — Everolimus was formulated as tablets of 5 mg strength. In both treatment arms, the study drug was given by continuous oral daily dosing of 10 mg (2 tablets x 5 mg) each morning.
  Other Names: RAD001
  Arms: Everolimus + BSC
Drug: Everolimus placebo — Placebo was formulated to be indistinguishable from the everolimus tablets, also formulated as tablets of 5 mg strength. In both treatment arms, the study drug was given by continuous oral daily dosing of 10 mg (2 tablets x 5 mg) each morning.
  Arms: Placebo + BSC
Drug: Best Supportive Care (BSC) — Best supportive care is defined as care in accordance with the local practice of an individual institution or center, specifically excluding anti-cancer treatments.

SUMMARY:
This study is designed to assess the safety and efficacy of RAD001 monotherapy in patients with advanced gastric cancer which has progressed after one or two lines of prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years old
* Histologically or cytologically confirmed and documented gastric adenocarcinoma
* Documented progression after 1 or 2 prior chemotherapy treatments for advanced disease
* ECOG Performance Status of < 2
* Lab parameters within specifically defined intervals
* Able to provide written informed consent

Exclusion Criteria:

* Patients who have received > 2 prior systemic therapies for advanced disease
* Administration of another anticancer therapy within 3 weeks prior to randomization
* Chronic treatment with steroids or another immunosuppressive agent
* Major surgery within 2 weeks prior to randomization
* Patients with CNS metastases
* Any other severe and/or uncontrolled medical condition

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2009-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (113):
- United States (8):
  - Highlands Oncology Group DeptofHighlandsOncologyGrp(2), Fayetteville, Arkansas
  - Loma Linda Oncology Medical Group Loma Linda, Redlands, California
  - Henry Ford Hospital Dept. of Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Texas Southwestern Medical Center DeptofSimmons Cancer Center(4), Dallas, Texas
  - The Center for Cancer and Blood Disorders Dept. of The Ctr for C & BD(2), Fort Worth, Texas
  - University of Texas/MD Anderson Cancer Center Gastrointestinal Med. Oncology, Houston, Texas
  - University of Washington Cancer Care Seattle Cancer Alliance, Seattle, Washington
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rio Negro, Viedma
- Australia (9):
  - Novartis Investigative Site, Canberra, Australian Capital Territory
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Kurralta Park, South Australia
  - Novartis Investigative Site, North Adelaide, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Footscray, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Prahran, Victoria
- Belgium (4):
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Canada (5):
  - Novartis Investigative Site, North Vancouver, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (11):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- France (15):
  - Novartis Investigative Site, Poitiers, France
  - Novartis Investigative Site, Avignon
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (8):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Mainz, Germany
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Offenburg
  - Novartis Investigative Site, Trier
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
- Italy (5):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Frattamaggiore
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sagamihara, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Utsunomiya, Tochigi
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Mitaka, Tokyo
- Mexico (2):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Mexico City, Mexico City
- Novartis Investigative Site, Amsterdam, Netherlands
- Novartis Investigative Site, Auckland, New Zealand
- Peru (2):
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- South Korea (4):
  - Novartis Investigative Site, Jeonju, Jeollabuk-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Taiwan (5):
  - Novartis Investigative Site, Niaosong Township, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
  - Novartis Investigative Site, Liouying Township
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla
- United Kingdom (6):
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, East Yorkshire
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] Ohtsu A, Ajani JA, Bai YX, Bang YJ, Chung HC, Pan HM, Sahmoud T, Shen L, Yeh KH, Chin K, Muro K, Kim YH, Ferry D, Tebbutt NC, Al-Batran SE, Smith H, Costantini C, Rizvi S, Lebwohl D, Van Cutsem E. Everolimus for previously treated advanced gastric cancer: results of the randomized, double-blind, phase III GRANITE-1 study. J Clin Oncol. 2013 Nov 1;31(31):3935-43. doi: 10.1200/JCO.2012.48.3552. Epub 2013 Sep 16. PMID 24043745
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com/etrials/searchTrial.do?trialID=717

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus 10mg/Daily: All patients were randomized to receive everolimus + BSC. All patients orally took two 5 mg tablets of everolimus once daily. Therefore, all patients in the everolimus arm took a total daily dose of 10 mg. Best supportive care was in accordance with the local practice of an individual institution or center, and specifically excluded anti-cancer treatments.
- Placebo: All patients were randomized to receive placebo + BSC. All patients orally took two 5 mg tablets of matching placebo once daily. Therefore, all patients in the placebo receive matching tablets of total daily dose of 10 mg. Best supportive care was in accordance with the local practice of an individual institution or center, and specifically excluded anti-cancer treatments.
Period: Overall Study
Arm/Group | Everolimus 10mg/Daily | Placebo
Started | 439 | 217
Discontinued Study Treatment | 428 | 217
Completed | 11 (Completed=Patients Still on Treatment; At data cutoff final analysis, 11 patients were on treatment) | 0
Not Completed | 428 | 217
Not completed — Adverse Event | 94 | 34
Not completed — Abnormal Laboratory Value | 1 | 0
Not completed — Withdrawal by Subject | 20 | 7
Not completed — Lost to Follow-up | 2 | 1
Not completed — Administrative Problems | 2 | 0
Not completed — Death | 16 | 5
Not completed — Disease Progression | 292 | 169
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus 10mg/Daily | Placebo | Total
Number analyzed (Participants) | 439 | 217 | 656
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.59) | 60.8 (11.61) | 60.4 (11.59)
Age, Customized [Number; unit: Participants]
  < 65 years | 260 | 129 | 389
  >=65 years | 179 | 88 | 267
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 56 | 173
  Male | 322 | 161 | 483
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 166 | 75 | 241
  Black | 3 | 1 | 4
  Asian | 251 | 126 | 377
  Native American | 0 | 1 | 1
  Other | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The primary objective of this study was to compare OS between everolimus + best supportive care (BSC) and placebo + BSC. OS, was defined as the time from date of randomization to the date of death due to any cause. If at the analysis cut-off date a patient was not known to have died, survival was censored at the date of the last contact. OS was analyzed using the Kaplan Meier estimates method.
Time Frame: 2.5 years
Population: The Full Analysis Set (FAS) consists of all randomized patients. Following the intent-to-treat principle, patients were analyzed according to the treatment and stratum that they were assigned to at randomization.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10mg/Daily | Placebo
Number analyzed (Participants) | 439 | 217
Months | 5.39 [4.80 to 6.01] | 4.34 [3.81 to 5.49]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival was defined as the time from the date of randomization to the date of the first documented disease progression or death due to any cause, where progression was based on Investigator assessment of baseline and post-baseline scans according to RECIST. Progression free survival was censored if no PFS event was observed before the first to occur out of (i) the cut-off date, or (ii) the date when a further anticancer therapy was started. The censoring date was the date of the last adequate tumor assessment before either of these two events occurred. If a PFS event was observed after two or more missing or non-evaluable tumor assessments, then the date of progression was censored at the date of the last adequate tumor assessment; for a PFS event observed after a single missing or non-evaluable tumor assessment, the actual date of disease progression was used. Anslsis was done using Kaplan-Meier estimates method.
Time Frame: 2.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10mg/Daily | Placebo
Number analyzed (Participants) | 439 | 217
Months | 1.68 [1.51 to 1.94] | 1.41 [1.38 to 1.45]

3. Secondary Outcome: Patient Reported Outcome (PRO): Time to Definitive Deterioration of European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire 30 (EORTC QLQ-C30) Scores
Description: The EORTC QLQ-C30 global health status/quality of life sub-scale (QL) was pre-specified as the primary domain of interest, followed by physical functioning (PF), social functioning (SF) and emotional functioning (EF).The EORTC QLQ-C30 questionnaire, along with a module specific for gastric cancer patients (EORTC QLQ-STO22), was used to evaluate PRO. The QLQ-C30 has five function scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and a global health status/quality of life scale. In addition, there are questions that assess specific symptoms. The QLQ-STO22 consists of 22 questions that make up five multi-item scales (dysphagia, pain, reflux, eating and anxiety) and four single-item scales (dry mouth, tasting, body image and hair loss).
Time Frame: 2.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10mg/Daily | Placebo
Number analyzed (Participants) | 439 | 217
Months
  In QL score by at least 5 % compared to baseline | 1.51 [1.28 to 1.84] | 1.45 [1.05 to 1.68]
  In PF score by at least 5 % compared to baseline | 1.35 [1.12 to 1.54] | 1.15 [1.02 to 1.64]
  In SF score by at least 5 % compared to baseline | 1.87 [1.84 to 2.30] | 1.87 [1.64 to 2.46]
  In EF score by at least 5 % compared to baseline | 1.84 [1.61 to 2.10] | 1.71 [1.41 to 1.87]

4. Secondary Outcome: Time to Definitive Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score
Description: The ECOG PS scale was used to classify patients according to their functional impairment, with scores ranging from 0 (fully active) to 5 (dead). An analysis of the time to definitive deterioration of the ECOG PS by one category of the score from baseline was performed. Definitive deterioration was defined as a definitive increase by one category from baseline in ECOG PS, with no later improvements observed during the course of the study. A single measure reporting an increase in ECOG PS is sufficient to consider it as a definitive worsening only if it was the last one available for the patient. Kaplan-Meier method was used to estimate the distribution function of time to definitive worsening.
Time Frame: 2.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus 10mg/Daily | Placebo
Number analyzed (Participants) | 439 | 217
Months | 2.30 [1.97 to 2.79] | 2.23 [1.87 to 2.92]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the proportion of patients with measurable disease in whom best overall response (OR) was either complete response (CR) or partial response (PR) according to RECIST criteria.
Time Frame: 2.5 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Everolimus 10mg/Daily | Placebo
Number analyzed (Participants) | 439 | 217
Participants
  Measurable Disease | 379 | 191
  Complete Response (CR) | 1 | 0
  Partial Response (PR) | 16 | 4
  Overall Response Rate (ORR) | 17 | 4

6. Secondary Outcome: Everolimus Steady State Concentraions at Predose (Cmin) and Cmax at Week 5
Description: Cmin is the minimum (trough) steady-state drug concentration in the blood during multiple dosing and Cmax is the maximum (peak) blood drug concentration after dose administration. Cmax is estimated as the maximum of C1h and C2H. C1h is 1 hour post-dose blood concentration and C2h is 2 hour post-dose blood concentration. Only valid pre-dose (Cmin), C1h, and C2h everolimus samples were included in the analysis. Valid pre-dose samples were confirmed blood samples collected at steady-state, collected immediately prior to dosing on the same study day, and collected at approximately 24 ± 4 hours after the previous dose and with no vomiting within the first 4 hours following the last dose. Valid C1h and C2h samples were confirmed blood samples collected at steady-state and within ± 1 hour window and with no vomiting within the first 4 hours following the current and previous dose.
Time Frame: Week 5
Population: PK analyses were based on the safety population in patients with evaluable samples. Only valid pre-dose (Cmin) & Cmax everolimus samples were included. For patients who were unable to tolerate the protocol-specified dosing schedule, dose adjustments were allowed to keep the patient on study drug. Some patients had dose reductions to 5mg daily.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Everolimus 5 mg/Day: Patients were randomized to receive everolimus + BSC. Patients orally took 1 5 mg tablet of everolimus once daily. Two of the 18 patients on the 5 mg arm, only had pre-dose evaluable samples.
Arm/Group | Everolimus 10mg/Daily | Everolimus 5 mg/Day
Number analyzed (Participants) | 218 | 18
ng/mL
  Pre-dose (Cmin) (n: 201,18) | 16.143 (10.7723) | 10.498 (6.1432)
  Cmax (n: 218,16) | 72.775 (36.5435) | 37.269 (27.2086)

7. Secondary Outcome: Everolimus Steady State Concentraions at Predose (Cmin) and Cmax by Region Asia vs. Rest of the World (ROW) at Week 5
Description: as for outcome 6
Time Frame: Week 5
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Everolimus 5mg/Day: Patients were randomized to receive everolimus + BSC. Patients orally took 5 mg tablet of everolimus once daily. One of the 11 patients on the 5 mg arm, only had a pre-dose evaluable sample.
Arm/Group | Everolimus 10mg/Daily | Everolimus 5mg/Day
Number analyzed (Participants) | 218 | 18
ng/mL
  Asia: Pre-dose (n:127, 11) | 16.804 (9.6163) | 9.921 (5.1565)
  Asia: Cmax (n:132, 10) | 73.568 (34.1898) | 34.580 (26.8110)
  Rest of the World: Pre-dose (n:74, 7) | 15.009 (12.5000) | 11.406 (7.8128)
  Rest of the World: Cmax (n:86, 6) | 71.558 (40.0655) | 41.750 (29.8074)

ADVERSE EVENTS:
Groups:
- Everolimus 10mg / Daily: Everolimus 10mg / daily
- Placebo: Placebo
Arm/Group | Everolimus 10mg / Daily | Placebo
Serious Adverse Events (participants affected / at risk) | 210/437 | 89/215
Other Adverse Events (participants affected / at risk) | 416/437 | 193/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10mg / Daily (N=437) | Placebo (N=215)
Anaemia (Blood and lymphatic system disorders) | 15 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 21 | 12
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 9 | 4
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 2 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 3
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 3
Ileus (Gastrointestinal disorders) | 5 | 0
Internal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 5 | 5
Intestinal perforation (Gastrointestinal disorders) | 3 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 9 | 9
Obstruction gastric (Gastrointestinal disorders) | 2 | 2
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Peritoneal disorder (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 3 | 1
Subileus (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 14 | 10
Asthenia (General disorders) | 12 | 6
Chest discomfort (General disorders) | 1 | 0
Device dislocation (General disorders) | 1 | 0
Device malfunction (General disorders) | 0 | 1
Device occlusion (General disorders) | 2 | 0
Drug intolerance (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 8 | 4
General physical health deterioration (General disorders) | 14 | 4
Hyperthermia (General disorders) | 2 | 0
Local swelling (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 10 | 1
Stent malfunction (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 2 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 5
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 0
Acinetobacter infection (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastric infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Lung infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 2 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 12 | 4
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic shock (Infections and infestations) | 4 | 0
Skin infection (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 0
Urosepsis (Infections and infestations) | 0 | 2
Colon injury (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Oesophageal injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
C-reactive protein increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 21 | 8
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 1
Fluid intake reduced (Metabolism and nutrition disorders) | 1 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Expressive language disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 4
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus 10mg / Daily (N=437) | Placebo (N=215)
Anaemia (Blood and lymphatic system disorders) | 108 | 42
Leukopenia (Blood and lymphatic system disorders) | 30 | 3
Neutropenia (Blood and lymphatic system disorders) | 47 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 77 | 4
Abdominal distension (Gastrointestinal disorders) | 39 | 20
Abdominal pain (Gastrointestinal disorders) | 90 | 49
Abdominal pain upper (Gastrointestinal disorders) | 51 | 26
Constipation (Gastrointestinal disorders) | 92 | 41
Diarrhoea (Gastrointestinal disorders) | 112 | 33
Dyspepsia (Gastrointestinal disorders) | 22 | 8
Nausea (Gastrointestinal disorders) | 129 | 63
Stomatitis (Gastrointestinal disorders) | 173 | 22
Vomiting (Gastrointestinal disorders) | 98 | 54
Asthenia (General disorders) | 67 | 18
Fatigue (General disorders) | 146 | 63
Oedema peripheral (General disorders) | 49 | 21
Pyrexia (General disorders) | 77 | 24
Alanine aminotransferase increased (Investigations) | 28 | 9
Aspartate aminotransferase increased (Investigations) | 34 | 8
Blood alkaline phosphatase increased (Investigations) | 34 | 6
Weight decreased (Investigations) | 87 | 19
Decreased appetite (Metabolism and nutrition disorders) | 202 | 76
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 25 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 52 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 46 | 16
Dizziness (Nervous system disorders) | 22 | 12
Dysgeusia (Nervous system disorders) | 26 | 7
Headache (Nervous system disorders) | 32 | 8
Insomnia (Psychiatric disorders) | 51 | 22
Proteinuria (Renal and urinary disorders) | 24 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 50 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 23 | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 22 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 9
Rash (Skin and subcutaneous tissue disorders) | 86 | 19

LIMITATIONS AND CAVEATS:
4 randomized patients, 2 patients each from the everolimus and placebo arms were excluded from the safety analyses as they did not receive any dose of study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.